CLINICAL TRIAL: NCT05966350
Title: Anti-Argonaute Antibodies for the Diagnosis of Sensory Neuronopathies
Acronym: AGO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN742021/CHUSTE
Record Dates: First submitted 2023-06-22; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-06

CONDITIONS: Autoimmune Diseases
Keywords: Sensory neuronopathy; Sensory ganglionopathy; Auto-antibody; Anti-AGO antibody
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum collection for anti-FGFR3 antibody studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sensory neuronopathies (SNN): Patients with Sensory neuronopathies (SNN) will be included.
  Interventions: Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 1; Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 2; Other: Comparison with Chi2 method; Other: Comparison of data with parametric Test (T-test); Other: Comparison of data with non-parametric test (ANNOVA)
- another peripheral neuropathy: Patients with small fiber neuropathy, chronic polyradiculoneuritis or other axonal neuropathy) will be included.
  Interventions: Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 1; Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 2; Other: Comparison with Chi2 method; Other: Comparison of data with parametric Test (T-test); Other: Comparison of data with non-parametric test (ANNOVA)
- dysimmune context without associated neuropathy.: Patient with dysimmune context without associated neuropathy will be included.
  Interventions: Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 1; Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 2; Other: Comparison with Chi2 method; Other: Comparison of data with parametric Test (T-test); Other: Comparison of data with non-parametric test (ANNOVA)

INTERVENTIONS:
Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 1 — Search of positivity with anti-AGO antibodies test
Diagnostic Test: Diagnosis of sensitive neuronopathy - phase 2 — Title of anti-AGO antibodies
Other: Comparison with Chi2 method — Clinical data from positive Argonaute (AGO) patients (age, sex, type of neuropathy, clinical manifestations of neuropathy, electroneuromyography , evolution of neuropathy, presence of associated autoimmune disease, response to possible immunomodulatory treatment) will be compared with those of negative patients using a Chi2 method for qualitative data.
Other: Comparison of data with parametric Test (T-test) — Clinical data from positive Argonaute (AGO) patients (age, sex, type of neuropathy, clinical manifestations of neuropathy, electroneuromyography, evolution of neuropathy, presence of associated autoimmune disease, response to possible immunomodulatory treatment) will be compared with those of negative patients using a parametric test (T-test).
Other: Comparison of data with non-parametric test (ANNOVA) — Clinical data from positive Argonaute (AGO) patients (age, sex, type of neuropathy, clinical manifestations of neuropathy, electroneuromyography , evolution of neuropathy, presence of associated autoimmune disease, response to possible immunomodulatory treatment) will be compared with those of negative patients using a non-parametric (ANNOVA).

SUMMARY:
Argonaute (AGO) proteins have been described as the target of antibodies in several autoimmune diseases including Sjögren Syndrome (SS). Sensory neuronopathies (SNN) are disorders affecting neurons in the dorsal root ganglia that may depend on an inflammatory process. However, identifying these cases needs the availability of specific biomarkers. The aim of this study is to test the prevalence of anti-AGO antibodies in a population of patients with Sensory neuronopathies (SNN) with and without associated autoimmune disease in comparison with other peripheral neuropathies to determine how anti-AGO antibodies may help the identification of potentially dysimmune Sensory neuronopathies (SNN).

DETAILED DESCRIPTION:
Sensory neuronopathies (SNN) are rare and debilitating diseases that fall under several etiologies. Among them, dysimmune forms are the most frequent but very difficult to identify when they do not occur in the context of associated systemic dysimmune disease (Sjögren Syndrome (SS) syndrome) because only a biopsy of the epiphytically unthinkable posterior spinal node would support the diagnosis. It is therefore necessary to have diagnostic biological markers of these forms to consider rapid treatment before irreversible neuronal degeneration.Using a protein-array technique, it has been showed that anti-FGFR3 antibodies was one of these markers and that it was associated with a clinical picture that differentiated from Sensory neuronopathies (SNN) without this antibody. Protein-array also allowed to identify another potentially interesting antibody for the diagnosis of Sensitive neuronopathies (NNS). This antibody recognizes the AGO1 protein. Anti-AGO1 antibodies have been described in association with system autoimmune diseases and in particular lupus but not in neurological diseases and more particularly in Sensory neuronopathies (SNN). The study want to validate the diagnostic interest of these antibodies by testing the collection of serums performed for studies on the anti-FGFR3 antibody and including patients with Sensory neuronopathies (SNN) and as controls of patients with another form of neuropathy and subjects with systemic autoimmune disease without peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sensory neuropathy

Exclusion Criteria:

* Patient not tested for anti-AGO antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sensory neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Sensitivity-specificity of Argonaute (AGO) antibodies for the diagnosis of sensory neuronopathies | 2 Years
  Sensitivity-specificity of Argonaute (AGO) antibodies screening

SECONDARY OUTCOMES:
Comparison of data between patients with anti-AGO antibodies versus patients without anti-AGO antibodies | 2 Years
  Clinical pattern of the neuropathy in patients with anti-AGO antibodies versus patients without anti-AGO antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ANTOINE, MDPHD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No